CLINICAL TRIAL: NCT01278082
Title: Double-blind, Randomised, Placebo-controlled, Multi-centre Phase III Clinical Study on the Efficacy and Tolerability of Budesonide Capsules Versus Placebo for Maintenance of Remission in Patients With Collagenous Colitis
Brief Title: SOIBD Collagenous Colitis Maintenance Study
Acronym: SCCMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Collaborators: The Swedish Organization for Studies on Inflammatory Bowel Disease (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUC-63/COC; 2007-001315-31 (EudraCT Number)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Induction and Maintaining Remission of Collagenous Colitis
Keywords: Randomized; double-blind; Placebo-controlled; budesonide; collagenous colitis; acute treatment; maintaining remission
MeSH Terms: conditions — Colitis, Collagenous | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Alternating daily dosing with 2 x 3 mg budesonide capsules OD and 1 x 3 mg budesonide capsule OD every second day
  Interventions: Drug: Budesonide
- B (Placebo Comparator): Alternating daily dosing with 2 placebo capsules OD and 1 placebo capsule OD every second day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — Alternating daily dosing with 2 x 3 mg budesonide capsules OD and 1 x 3 mg budesonide capsule OD every second day
  Other Names: Budenofalk 3mg capsules
  Arms: A
Drug: Placebo — Alternating daily dosing with 2 placebo capsules OD and 1 placebo capsule OD every second day.
  Arms: B

SUMMARY:
This study aims to demonstrate the superiority of budesonide compared to placebo as maintenance therapy in keeping patients in remission over a one-year period

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent,
2. Patients aged >= 18 years,
3. Histologically established diagnosis of collagenous colitis (CC) defined as:

   1. Thickened sub-epithelial collagen layer >= 10 µm on well-orientated sections,
   2. Increased amount of inflammatory cells indicating chronic inflammation in the lamina propria,
4. History of non-bloody, watery diarrhoea for more than 2 weeks prior screening in patients with newly diagnosed collagenous colitis, or history of clinical relapse for more than 1 week prior screening in patients with previously established collagenous colitis,
5. A mean of >= 3 stools/day, thereof a mean of >= 1 watery stools/day, during the week prior baseline,
6. Women of child-bearing potential and being heterosexually active have to apply appropriate contraceptive methods, e.g., hormonal contraception, intrauterine device (IUD), double-barrier method of contraception (e.g., use of a condom and spermicide), or partner has undergone vasectomy. The investigator is responsible for determining whether the subject has adequate birth control for study participation.

Exclusion Criteria:

1. Other significant abnormalities at colonoscopy that may have been the cause of diarrhoea, with the exception of colonic diverticulosis and polyps < 2 cm,
2. Infectious cause of diarrhoea,
3. Untreated active celiac disease,
4. Clinical suspicion of drug-induced collagenous colitis,
5. Any severe concomitant cardiovascular, renal, endocrine, or psychiatric disorder,
6. Abnormal hepatic function (ALT or ALP > 2.5 x upper limit of normal [ULN]), liver cirrhosis, or portal hypertension,
7. Local intestinal infection,
8. Radiation therapy towards the abdominal or pelvic region,
9. Diabetes mellitus, infection, glaucoma, tuberculosis, peptic ulcer disease, or hypertension if careful medical monitoring is not ensured,
10. Known established cataract,
11. Known hereditary problems of galactose or fructose intolerance, glucose-galactose malabsorption, sucrase-isomaltase insufficiency, Lapp lactase deficiency, or congenital lactase deficiency,
12. Established osteoporosis with T-score < -2.5,
13. Pregnancy or lactation,
14. History of cancer in the last five years,
15. History of significant bowel resection,
16. Therapy with immunomodulators (azathioprine, 6-mercaptopurine, or methotrexate) in the last 3 months,
17. Treatment with oral, rectal, or intravenous corticosteroids including budesonide in the last month,
18. Known intolerance/hypersensitivity to study drug or drugs of similar chemical structure or pharmacological profile,
19. Patients who are unable to adhere to the study visit schedule and other protocol requirements according to the judgement of the investigator,
20. Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-04; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients being in remission over 52 weeks. | 52 weeks
  Remission is defined as a mean of < 3 stools/day, thereof a mean of < 1 watery stools/day

SECONDARY OUTCOMES:
Proportion of patients in remission at wk 4, 13, 26, and 39. | 39 weeks
  Remission is defined as a mean of < 3 stools/day, thereof a mean of < 1 watery stools/day
Adverse events (AEs) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Müller, Dr, Study Director — Dr. Falk Pharma GmbH
Locations (2):
- Center of digestive diseases, Hamburg, Germany
- University Hospital of Linköping, Linköping, Sweden

REFERENCES:
- [Result] Munch A, Bohr J, Miehlke S, Benoni C, Olesen M, Ost A, Strandberg L, Hellstrom PM, Hertervig E, Armerding P, Stehlik J, Lindberg G, Bjork J, Lapidus A, Lofberg R, Bonderup O, Avnstrom S, Rossle M, Dilger K, Mueller R, Greinwald R, Tysk C, Strom M; BUC-63 investigators. Low-dose budesonide for maintenance of clinical remission in collagenous colitis: a randomised, placebo-controlled, 12-month trial. Gut. 2016 Jan;65(1):47-56. doi: 10.1136/gutjnl-2014-308363. Epub 2014 Nov 25. PMID 25425655